CLINICAL TRIAL: NCT00030862
Title: Phase II Single-Arm Trial Of CPT-11 (Irinotecan HC1; Camptosar Injection)/Cisplatin In Patients With Advanced Esophageal Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Locally Advanced or Metastatic Cancer of the Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 01-123; CDR0000069204 (Registry Identifier: PDQ (Physician Data Query)); PHARMACIA-440E-ONC-0020-319; NCI-G01-2050
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Esophageal Cancer
Keywords: stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; squamous cell carcinoma of the esophagus; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Adenocarcinoma Of Esophagus | interventions — Cisplatin; Irinotecan

INTERVENTIONS:
Drug: cisplatin
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining irinotecan and cisplatin in treating patients who have locally advanced unresectable or metastatic cancer of the esophagus that has not been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective tumor response rate in patients with previously untreated locally advanced unresectable or metastatic esophageal cancer treated with irinotecan and cisplatin.
* Determine the dysphagia relief in patients treated with this regimen.
* Determine the time to progression and overall survival of patients treated with this regimen.
* Determine the safety of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive cisplatin IV over 1-2 hours and irinotecan IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma or adenocarcinoma of the esophagus

  * Previously untreated
  * Locally advanced unresectable or metastatic disease
  * More than 50% of tumor must involve esophagus or gastroesophageal (GE) junction if tumor extends below the GE junction into the proximal stomach
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR
  * At least 10 mm by spiral CT scan
  * The following are not considered measurable disease:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusions
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
    * Tumor lesions in previously irradiated areas
* No carcinomatous meningitis or untreated brain metastases

  * Brain metastases allowed if asymptomatic and patient is on stable or tapering dose of steroids
* Large pleural effusions must have been previously drained and sclerosed or otherwise controlled

  * Small, stable, asymptomatic pleural effusions allowed
* Dysphagia allowed

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* AST no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* No known Gilbert's disease

Renal:

* Creatinine no greater than 1.5 mg/dL
* Calcium less than 12.0 mg/dL

Cardiovascular:

* No history of significant cardiovascular disease
* No inadequately controlled hypertension
* No unstable angina
* No myocardial infarction within the past 6 months
* No ventricular cardiac arrhythmias requiring medication
* No history or treatment for congestive heart failure

Pulmonary:

* No interstitial pneumonia
* No fibroid lung

Other:

* No serious active infection
* No uncontrolled diabetes mellitus (random blood sugar at least 300 mg)
* No peripheral neuropathy grade 2 or greater
* No other malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or any other malignancy that does not carry a worse prognosis than advanced esophageal cancer
* No other serious underlying medical condition that would preclude study
* No other concurrent disease that would preclude study
* No psychiatric illness or other significant mental impairment that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics
* At least 2 weeks since prior radiotherapy and recovered
* No prior radiotherapy to the pelvis

Surgery:

* See Disease Characteristics
* Not specified

Other:

* No concurrent phenytoin or phenobarbital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Ilson, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States